CLINICAL TRIAL: NCT02916771
Title: Phase II Trial of Combination of Ixazomib and Lenalidomide and Dexamethasone in Smoldering Multiple Myeloma
Brief Title: Trial of Combination of Ixazomib and Lenalidomide and Dexamethasone in Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celgene (Industry); Takeda (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Irene M. Ghobrial, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-313
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixazomib (Experimental): * Cycles 1-9
    * Ixazomib is administered orally on days 1, 8, 15 on a 28 days cycle
    * Lenalidomide is administered orally on days 1-21 on a 28 days cycle
    * Dexamethasone is administered orally on days 1, 8, 15, 22 on a 28 days cycle
  * Cycle 10-24
    * Ixazomib is administered orally on days 1, 8, 15 on a 28 days cycle
    * Lenalidomide is administered orally on days 1-21 on a 28 days cycle
  * Supportive measures consistent with optimal patient care may be given throughout the study
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Oral, proteasome inhibitor
  Other Names: Ninlaro
Drug: Lenalidomide — Oral, immunomodulatory agent
  Other Names: Revlimid
Drug: Dexamethasone — Oral, steroid
  Other Names: Decadron

SUMMARY:
This research study is evaluating a new drug called "ixazomib" as a possible treatment for Smoldering Multiple Myeloma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial, which tests the effectiveness of an investigational drug(s). The investigational drugs used in this research study are Ixazomib, Lenalidomide and Dexamethasone.

"Investigational" means that the FDA (the U.S. Food and Drug Administration) has not approved the combination of Ixazomib, Lenalidomide and Dexamethasone as a treatment regimen for Smoldering Multiple Myeloma. The purpose of this research study is to learn whether the combination of Ixazomib, Lenalidomide, and Dexamethasone works in treating Smoldering Multiple Myeloma.

Ixazomib is a drug that may kill or stop cancer cells from growing by blocking the proteasome within the cell, which is responsible for degrading or breaking down a variety of proteins. This type of drug is called a proteasome inhibitor. Lenalidomide is an immunomodulatory drug, meaning it modifies the participant immune system to help fight the participant disease. Dexamethasone is a steroid, which is usually combined with other drugs to enhance their effects to fight the participant disease.

Ixazomib is approved by the FDA in combination with Lenalidomide and Dexamethasone for the treatment of Multiple Myeloma and is currently being evaluated for use in the treatment of several types of cancers. Both Lenalidomide and Dexamethasone have been previously approved by the FDA for the treatment of Multiple Myeloma, as well as several other cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Must meet criteria of high risk smoldering MM based on the criteria described below:
* Definition of high-risk SMM:

  --Bone marrow clonal plasma cells ≥10% and ≤60% and any one or more of the following:
  * Serum M protein ≥3.0g/dL (IgA, IgG, IgM, or IgD)
  * IgA SMM
  * Immunoparesis with reduction of two uninvolved immunoglobulin isotypes
  * Serum involved/uninvolved free light chain ratio ≥8 (but less than 100)

    ----Free Light Chain Smoldering Myeloma patients as defined in section 2.4 are not excluded
  * Progressive increase in M protein level (Evolving type of SMM)

    ----Increase in serum monoclonal protein by ≥10% on two successive evaluations within a 6 month period
  * Bone marrow clonal plasma cells 50-60%
  * Abnormal plasma cell immunophenotype (≥95% of bone marrow plasma cells are clonal) and reduction of one or more uninvolved immunoglobulin isotypes
  * t (4;14) or del 17p or 1q gain
  * Increased circulating plasma cells
  * MRI with diffuse abnormalities or 1 focal lesion
  * PET-CT with one focal lesion with increased uptake without underlying osteolytic bone destruction
  * Urine monoclonal light chain excretion ≥500 mg/24 hours
* ECOG Performance Status (PS) 0, 1, or 2 (Appendix A)
* The following laboratory values obtained ≤ 21 days prior to registration and confirmed prior to the first dose of study drug:

  * ANC ≥ 1000/uL
  * PLT ≥ 75,000/uL. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
  * Total bilirubin ≤ 1.5 mg/dL (If total is elevated check direct and if normal patient is eligible.)
  * AST ≤ 3 x institutional upper limit of normal (ULN)
  * ALT ≤ 3 x institutional upper limit of normal (ULN)
  * Calculated creatinine clearance ≥ 30 mL/min
* Ability to understand and the willingness to sign a written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female patients who are postmenopausal for at least 1 year before the screening visit or are surgically sterile. Females of childbearing potential* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS®) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. Female patients must agree to practice two effective methods of birth control from the time of signing the informed consent form though 90 days after the last dose of study drug
* A female of childbearing potential is a sexually mature female who:

  * Has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or
  * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy during the entire study treatment period and through 90 days after the last dose of study drug OR agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* No evidence of CRAB* criteria or new criteria of active MM which including the following:

  * Increased calcium levels (corrected serum calcium >0.25 mmol/dL above the upper limit of normal or >.275 mmol/dL) related to MM
  * Renal insufficiency (attributable to MM)
  * Anemia (Hb 2g/dL below the lower limit of normal or <10g/dL) related to MM
  * Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
  * Bone marrow plasma cells ≥60%
  * Serum involved/uninvolved FLC ratio ≥100, provided the absolute level of the involved free light chain is at least 100 mg/L and repeated twice
  * MRI with two or more focal lesion that is at least 5 mm or greater in size
* Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational. Prior therapy with bisphosphonate is allowed. Prior radiation therapy to a solitary plasmacytoma is allowed.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women will be excluded from the study because lenalidomide is an agent with the potential for teratogenic or abortifacient effects.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ixazomib or lenalidomide.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Major surgery within 14 days before enrollment.
* Known Amyloid involvement.
* Myeloma-related central nervous system involvement.
* Systemic treatment, within 14 days before the first dose of ixazomib with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Grade 2 peripheral neuropathy or higher or grade 1 with pain on clinical examination during the screening period.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
* Previous treatment with ixazomib, or participation in a study with ixazomib whether treated with ixazomib or not.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nadeem O, Aranha MP, Redd R, Timonian M, Magidson S, Lightbody ED, Alberge JB, Bertamini L, Dutta AK, El-Khoury H, Bustoros M, Laubach JP, Bianchi G, O'Donnell E, Wu T, Tsuji J, Anderson KC, Getz G, Trippa L, Richardson PG, Sklavenitis-Pistofidis R, Ghobrial IM. Deeper response predicts better outcomes in high-risk-smoldering-myeloma: results of the I-PRISM phase II clinical trial. Nat Commun. 2025 Jan 3;16(1):358. doi: 10.1038/s41467-024-55308-5. PMID 39753553
- [Derived] Nadeem O, Aranha MP, Redd R, Timonian M, Magidson S, Lightbody ED, Alberge JB, Bertamini L, Dutta AK, El-Khoury H, Bustoros M, Laubach JP, Bianchi G, O'Donnell E, Wu T, Tsuji J, Anderson K, Getz G, Trippa L, Richardson PG, Sklavenitis-Pistofidis R, Ghobrial IM. Long-Term Follow-Up Defines the Population That Benefits from Early Interception in a High-Risk Smoldering Multiple Myeloma Clinical Trial Using the Combination of Ixazomib, Lenalidomide, and Dexamethasone. medRxiv [Preprint]. 2024 Apr 19:2024.04.19.24306082. doi: 10.1101/2024.04.19.24306082. PMID 38699307

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixazomib: * Cycles 1-9
    * Ixazomib is administered orally on days 1, 8, 15 on a 28 days cycle
    * Lenalidomide is administered orally on days 1-21 on a 28 days cycle
    * Dexamethasone is administered orally on days 1, 8, 15, 22 on a 28 days cycle
  * Cycle 10-24
    * Ixazomib is administered orally on days 1, 8, 15 on a 28 days cycle
    * Lenalidomide is administered orally on days 1-21 on a 28 days cycle
  * Supportive measures consistent with optimal patient care may be given throughout the study
  Ixazomib: Oral, proteasome inhibitor
  Lenalidomide: Oral, immunomodulatory agent
  Dexamethasone: Oral, steroid
Period: Overall Study
Arm/Group | Ixazomib
Started | 61
Completed | 50
Not Completed | 11
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 1
Not completed — Began treatment for another active malignancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 64 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Proportion Of High Risk SMM Patients Who Are Progression Free 2 Years After Receiving IRD Combination Therapy
Description: The proportion of patients who achieve progression free at 2 years will be compared to the rate published for the high risk SMM. By the Mayo Clinic model for risk factors, the median time to progression for patients with high risk SMM was only 1.9 years. Therefore, we assume that, a 2-years progression-free rate of 50% will not be considered promising and a true progression free rate of 75% or higher will be considered promising.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 55
Participants | 50

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival is defined as the time from protocol therapy initiation to the disease progression or death from any cause, censored at date last known progression free for those who have not progressed or died
Time Frame: Time from protocol therapy initiation to the disease progression or death from any cause, censored at date last known progression free for those who have not progressed or died, or up to 60 months post initiation of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 53
Participants | 52

3. Secondary Outcome: Time To Progression
Description: Time to progression (TTP) is defined as the time from protocol therapy initiation until documented progression, censored at date last known progression-free for those who have not progressed.
Time Frame: The time from protocol therapy initiation until documented progression, censored at date last known progression-free for those who have not progressed or up to 60 months post initiation of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 55
months | 49.9 [39.9 to NA] — Not reached

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from objective response to disease progression or death, or date last known progression-free and alive for those who have not progressed or died
Time Frame: time from objective response to disease progression or death, or date last known progression-free and alive for those who have not progressed or died, or up to 60 months post initiation of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib
Number analyzed (Participants) | 51
months | 47.4 [37 to NA] — Not reached

5. Secondary Outcome: Objective Response Rate
Description: The objective response rate is defined as partial response or better according to the modified IMWG criteria.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 55
Participants | 51

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from protocol therapy initiation to death or date last known alive
Time Frame: Time from protocol therapy initiation to death or date last known alive, or up to 60 months post initiation of treatment
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Ixazomib
Number analyzed (Participants) | 55
years | NA [NA to NA] — Median overall survival was not reached at study completion.

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from the time of signing informed consent, through 30 days after administration of the last dose of study drug (approximately 2 years). Deaths were assessed for up to 60 months post initiation of treatment.
Arm/Group | Ixazomib
All-Cause Mortality (participants affected / at risk) | 1/55
Serious Adverse Events (participants affected / at risk) | 15/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=55)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung infection (Infections and infestations) | 2
Allergic reaction (Immune system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Skin infection (Infections and infestations) | 1
Dehdyration (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Neutrophil count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Platelet count decreased (Investigations) | 1
Respiratory, thoracic and mediastinal disorders- Other (Respiratory, thoracic and mediastinal disorders) | 2 — COVID-19
Syncope (Nervous system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Upper respiratory infection (Infections and infestations) | 1 — RSV
Cognitive disturbance (Nervous system disorders) | 1
Infections and infestations- Other (Infections and infestations) | 1 — Influenza A
Intracranial hemorrhage (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Psychiatric disorders - Other (Psychiatric disorders) | 1 — Intentional overdose
Depression (Psychiatric disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Atrial fibrillation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=55)
White blood cell decreased (Investigations) | 44
Neutrophil count decreased (Investigations) | 43
Fatigue (General disorders) | 41
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 38
Diarrhea (Gastrointestinal disorders) | 37
Anemia (Blood and lymphatic system disorders) | 33
Nausea (Gastrointestinal disorders) | 33
Platelet count decreased (Investigations) | 33
Edema limbs (General disorders) | 31
Insomnia (Psychiatric disorders) | 31
Peripheral sensory neuropathy (Nervous system disorders) | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 27
Constipation (Gastrointestinal disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Dizziness (Nervous system disorders) | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21
Headache (Nervous system disorders) | 19
Upper respiratory infection (Infections and infestations) | 18
Vomiting (Gastrointestinal disorders) | 18
Dysgeusia (Nervous system disorders) | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Lymphocyte count decreased (Investigations) | 15
Alanine aminotransferase increased (Investigations) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Blurred vision (Eye disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 13
Flushing (Vascular disorders) | 12
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12
Bruising (Injury, poisoning and procedural complications) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 11
Fever (General disorders) | 11
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11
Hypertension (Vascular disorders) | 11
Tremor (Nervous system disorders) | 11
Bloating (Gastrointestinal disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 10
Aspartate aminotransferase increased (Investigations) | 9
Irritability (General disorders) | 9
Cognitive disturbance (Nervous system disorders) | 8
Sinus bradycardia (Cardiac disorders) | 8
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7
Blood bilirubin increased (Investigations) | 7
Dry mouth (Gastrointestinal disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 7
Pain (General disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Hot flashes (Vascular disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6
Concentration impairment (Nervous system disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 5
Flu like symptoms (General disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 5
Localized edema (General disorders) | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5
Urinary tract infection (Infections and infestations) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Agitation (Psychiatric disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Bronchial infection (Infections and infestations) | 4
Chills (General disorders) | 4
Depression (Psychiatric disorders) | 4
Dry eye (Eye disorders) | 4
Edema face (General disorders) | 4
Eye disorders - Other (Eye disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Lung infection (Infections and infestations) | 4
Memory impairment (Nervous system disorders) | 4
Nervous system disorders - Other (Nervous system disorders) | 4
Palpitations (Cardiac disorders) | 4
Restlessness (Psychiatric disorders) | 4
Rhinitis inefective (Infections and infestations) | 4
Sinus pain (Nervous system disorders) | 4
Skin atrophy (Skin and subcutaneous tissue disorders) | 4
Weight loss (Investigations) | 4
Atrial fibrilation (Cardiac disorders) | 3
Ear pain (Ear and labyrinth disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Presyncope (Nervous system disorders) | 3
Renal and urinary disorders- Other (Renal and urinary disorders) | 3
Sinusitis (Infections and infestations) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Skin infection (Infections and infestations) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT02916771/Prot_SAP_000.pdf